CLINICAL TRIAL: NCT00006023
Title: Master Protocol for Metastatic Hormone-Resistant Prostatic Carcinoma - Phase II Trials - Protocol 5: Capecitabine
Brief Title: Capecitabine in Treating Patients With Metastatic Prostate Cancer That Has Not Responded to Hormone Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: SAKK 08/00; SWS-SAKK-08/00 (Other: SAKK); EU-20020 (Other: EU)
Record Dates: First submitted 2000-07-05; First posted 2004-03-24 (Estimated); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Prostate Cancer
Keywords: stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: capecitabine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of capecitabine in treating patients who have metastatic prostate cancer that has not responded to hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy of capecitabine in terms of PSA response, PSA response duration, and time to PSA progression in patients with metastatic hormone refractory prostate cancer. II. Evaluate the toxicity of this treatment in these patients. III. Evaluate the correlation between PSA response and quality of life in these patients.

OUTLINE: This is a multicenter study. Patients receive oral capecitabine twice daily on days 1-14. Treatment continues every 21 days for up to 8 courses in the absence of disease progression or unacceptable toxicity. Quality of life is assessed on days 1 and 8 of the first course of treatment, on day 1 of each course thereafter, and at treatment failure. Patients are followed every 3 months until disease progression.

PROJECTED ACCRUAL: A total of 14-25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed metastatic hormone refractory prostate cancer Disease progression after orchiectomy or during hormonal therapy Measurable or evaluable disease At least 2 consecutive increases in PSA At least 1 week between reference value and first increase OR Third value must be higher than second if second value is less than reference value PSA at least 5 ng/mL No leptomeningeal or brain metastases

PATIENT CHARACTERISTICS: Age: 18 to 85 Performance status: WHO 0-2 Life expectancy: Not specified Hematopoietic: WBC at least 3,500/mm3 OR Granulocyte count at least 2,000/mm3 Hemoglobin at least 9.0 g/dL Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) SGOT no greater than 2.5 times ULN Renal: Creatinine no greater than 1.5 times ULN Other: No other prior malignancies in past 5 years except curatively treated basal cell or squamous cell carcinoma of the skin No other significant disease that would preclude study No concurrent active severe infections

PRIOR CONCURRENT THERAPY: Biologic therapy: Prior gene therapy and antibody therapy allowed Chemotherapy: No prior cytostatic chemotherapy, including estramustine Endocrine therapy: See Disease Characteristics At least 1 month since prior antiandrogen therapy (e.g., flutamide or bicalutamide) without tumor response OR Concurrent antiandrogen therapy allowed if clinically unacceptable to discontinue use If disease progressed while receiving hormonal agents (e.g., goserelin, leuprolide, diethylstilbestrol), therapy must continue during study Radiotherapy: At least 4 weeks since prior radiotherapy No prior radiotherapy to lesions to be evaluated No concurrent radiotherapy to more than one area Surgery: See Disease Characteristics Other: Prior noncytostatic therapy allowed At least 1 month since prior investigational drugs

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-03; Primary Completion 2001-06 (Actual); Study Completion 2001-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rudolf Morant, MD, Study Chair — Cantonal Hospital of St. Gallen
Locations (2):
- Switzerland (2):
  - Spitalzentrum Biel, Biel
  - Kantonsspital - Saint Gallen, Sankt Gallen

REFERENCES:
- [Result] Morant R, Bernhard J, Dietrich D, Gillessen S, Bonomo M, Borner M, Bauer J, Cerny T, Rochlitz C, Wernli M, Gschwend A, Hanselmann S, Hering F, Schmid HP. Capecitabine in hormone-resistant metastatic prostatic carcinoma - a phase II trial. Br J Cancer. 2004 Apr 5;90(7):1312-7. doi: 10.1038/sj.bjc.6601673. PMID 15054447